CLINICAL TRIAL: NCT06536426
Title: Effectiveness of a Knee Isometric Program on Reducing Anterior Knee Pain and Improving Functional Outcomes
Brief Title: Knee Isometric Program (KIP) Home Exercise Programs (HEP) Physical Therapy (PT) Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was determined to be too difficult to run following the enrollment of a few participants over the course of a year. No preliminary or final results were obtained.
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, John S. Dunn Chair in Orthopedic Surgery, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037838
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee Isometric Program (KIP) - Intervention (Experimental): This group will incorporate the KIP protocol, which is a modified physical therapy regimen that is less time-intensive than the gold standard counterpart. Typical structured/skilled physical therapy occurs over the course of 4-8 weeks with 1-2 visits per week to establish improved lower extremity muscle strength, education, and improve gross function. Home exercise programs (HEP) are utilized in tandem with physical therapy visits so that patients are completing interventions 4-5 days per week. Long-term maintenance is generally provided via a refined comprehensive HEP on completion and discharge from formal physical therapy.
  Interventions: Behavioral: Knee Isometric Program (KIP)
- Patellofemoral Clinical Practice Guideline (CPG) - Control (No Intervention): This group will incorporate the standard of care physical therapy regimen which includes a specific and structured combination of quadriceps and gluteal strengthening as defined in the patellofemoral pain clinical practice guideline. Typical structured/skilled physical therapy occurs over the course of 4-8 weeks with 1-2 visits per week to establish improved lower extremity muscle strength, education, and improve gross function. Home exercise programs (HEP) are utilized in tandem with physical therapy visits so that patients are completing interventions 4-5 days per week. Long-term maintenance is generally provided via a refined comprehensive HEP on completion and discharge from formal physical therapy.

INTERVENTIONS:
Behavioral: Knee Isometric Program (KIP) — The KIP physical therapy protocol follows the schedule outlined below:
  * Session 1 (Completed 4-5 days/week including HEP): Double Leg wall sit 3x30 seconds, Double Leg glute bridge hold 3x30 seconds, Single Leg Stance hold 3x1 minutes, Lunge hold 3x1 minutes
  * Session 2 (Completed 4-5 days/week including HEP): Single Leg wall sit 3x20 seconds, Single Leg glute bridge hold 3x20 seconds, Single Leg stance hold 2x1.5 minutes, Lunge hold 2x1.5 minutes
  * Session 3 (Completed 4-5 days/week including HEP): Single leg wall sit 3x40 seconds, Single leg glute bridge hold 3x40 seconds, Single leg stance hold 2x3 minutes, Lunge hold 2x3 minutes
  * Session 4 (Completed 4-5 days/week including HEP): Single leg wall sit 3x40 seconds, Single leg glute bridge hold 3x40 seconds, Single leg stance hold 2x3 minutes, Lunge hold 2x3 minutes
  Arms: Knee Isometric Program (KIP) - Intervention

SUMMARY:
The purpose of this study is to evaluate the efficacy of a knee isometric program (KIP) as compared to the current gold standard treatment for anterior knee pain (Patellofemoral Clinical Practice Guideline [CPG] - Academy of Orthopedic Physical Therapy).

DETAILED DESCRIPTION:
Participants will be randomly allocated into the KIP or control intervention via spreadsheet randomization algorithm at the time of consenting. Each patient will have equivalent experiences for the duration of the study regardless of allocation. Time spent with the physical therapist, daily length of exercise program, outcome measures recorded, and home education materials will all be similar for each group. Participants will be asked to refrain from any outside forms of lower extremity strengthening or training. Usage of pain medication (including over-the-counter and prescription drugs) will be documented in the pain journal. Proper use of the pain journal will be explained during consent and again at the initial intake session.

ELIGIBILITY:
Inclusion Criteria:

* Accept all provisions of the study and agree to complete the program in its entirety
* Age between 18-65
* Complaint of anterior knee pain for at least 4 weeks, but no more than 12 months
* Prescribed referral for physical therapy for their knee(s) from one of the investigators

Exclusion Criteria:

* Potential participant does not agree to comply with study protocols or does not wish to be subjected to a random group allocation
* Any neurological or degenerative musculoskeletal condition involving the lower extremities
* Ages outside of 18-65
* Surgical history or fracture within the last 12 months on the affected extremity(ies)
* Currently participating in a structured strength training program
* Inability to access clinic for data collection or follow-up sessions
* Significant anatomical anomaly or limb alignment disorder as diagnosed by medical professional (femoral anteversion/retroversion, patella alta/baja, varus/valgus deformities, patella deformities/fractures, osteotomy procedures, limb lengthening procedures)
* Significant cartilage damage as diagnosed by medical professional (grade 3+ chondral defects of the femur or patella)
* Any other condition that limits full weight bearing of the affected lower extremity(ies)
* Vulnerable populations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Subjective Pain | Baseline, 2 weeks, 4 weeks, 6 weeks, 12 weeks
  Participants will complete the Numerical Pain Rating Scale (NPRS) in a pain and medication journal in order to subjectively rate their pain over over 4-5 days between each session, except for after session 4 in which they will document twice a day for 20 days. The NPRS rates pain on a scale of 0 to 10 with 0 being no pain and 10 being the worst pain imaginable, and subjects will reflect pain pre and post physical therapy. Additionally, they will be asked to reflect any pain medication that they take on a given day.
Knee Function | Baseline, 12 weeks
  Participants will complete the lower extremity functional scale (LEFS) at session 1 and at session 5 (one month follow up visit after completing physical therapy) in order to determine any change in knee function across those time periods. The LEFS is a 20 question survey that asks about a person's ability to perform everyday tasks and each question is scored on a scale from 0 to 4 with 0 being extreme difficulty or unable to perform activity and 4 being no difficulty. These responses are then summed to get a total score out of 80 maximum points, and the lower the score, the greater the disability.
Objective Muscular Strength Performance | Baseline, 12 weeks
  Participants will have their quad strength measured using a handheld dynamometer (HHD) at session 1 and session 5 of their study visits in order to determine with that data how muscular strength changes following each physical therapy regimen.
Functional Stability | Baseline, 12 weeks
  Functional stability will be assessed at sessions 1 and 5 to determine each participant's dynamic balance, and it will be used to assess anterior reach specifically. This test has the participant stand on one leg while reaching out in 3 different directions with the other lower extremity, and thus measures strength, stability, and balance in multiple directions. The composite score is calculated by summing the three reach directions. Higher scores reflect better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No